CLINICAL TRIAL: NCT01429740
Title: A Phase 1, Placebo-Controlled, Randomized, Subject- And Investigator-Blind, Sponsor-Open, Crossover Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PF-05180999 After First-Time Administration Of Single Ascending Doses To Healthy Adult Subjects
Brief Title: A Study Of The Safety, Tolerability And Pharmacokinetics Of Single Doses Of PF-05180999 In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B3441001
Record Dates: First submitted 2011-08-24; First posted 2011-09-07 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: PF 05180999; safety; pharmacokinetics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05180999 (Experimental)
  Interventions: Drug: PF-05180999
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05180999 — Ascending single oral doses of 0.1, 0.3, 1.0, 3, 10, 30, 100, and 250 mg oral solution or capsules
  Arms: PF-05180999
Drug: Placebo — Placebo oral solution or capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of 14 days of treatment with PF-05180999 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

male or female of non-childbearing potential,

Exclusion Criteria:

Evidence of clinically significant medical illness, history of seizures, any condition possibly affecting drug absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Composite (or profile) of Pharmacokinetics | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose on Day 1 and Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3441001&StudyName=A%20Study%20Of%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20Single%20Doses%20Of%20PF-05180999%20In%20Healthy%20Adults